CLINICAL TRIAL: NCT02463292
Title: Quality of Life, Psychological Adjustment and Academic Achievement in Young Adults With Congenital Heart Disease
Brief Title: Quality of Life in Young Adults With Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Principal Investigator, Markus A. Landolt, Prof. Markus Landolt, PhD, University Children's Hospital, Zurich
Other Study IDs: QLYACHD
Record Dates: First submitted 2015-05-28; First posted 2015-06-04 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Congenital Heart Disease
Keywords: quality of life; young adults; congenital heart disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patient group: The patient group will consist of a maximum of 350 patients (male and female subjects,18 years to 30 years of age, in command of the German language)) with congenital heart disease (Tetralogy of Fallot, Transposition of the great arteries, univentricular heart disease, ventricular septal defect) treated at the cardiologic department of the University Hospital Zurich. Eligible patients will be contacted by the study nurse during the outpatient consultation at the university hospital. No intervention.
  Interventions: Other: no intervention
- peer control group: The control group will be recruited as good friends (same gender, approx. same age of the patients, in command of the German language). The patients will be given a study information for controls to hand this to their good friend and ask the friend to contact the study nurse for participation in the study. No intervention.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This study aims to evaluate the psychosocial situation of adult congenital heart disease (CHD) patients in terms of health-related quality of life, mental health, academic achievement, and employment status. By assessing a wide variety of medical (e.g., disease severity) and psychosocial (e.g., life events, coping strategies, personality) risk factors it will be possible to better understand the variables that influence psychosocial outcome of young adults with congenital heart disease. This will further improve the understanding of the lifelong consequences of a congenital heart malformation. Factors that proof to be predictors of favorable outcome represent a resource of resilience and therefore should play an important role in the care of CHD patients. By implementing those results in patient care the investigators aim to achieve an improved psychosocial outcome among adult congenital heart disease (ACHD).

Hypothesis 1: It is expected that perceived health status, health-related quality of life and psychological adjustment will not differ between the patient and the control group. However, academic achievement and employment status are expected to be poorer in young adults with congenital heart disease compared to healthy controls.

Hypothesis 2: It is assumed that parental socioeconomic status, problems in emotional regulation and impaired social support will be related to a negative psychosocial outcome and health-related quality of life. Moreover, the investigators hypothesize that disease severity is associated with academic outcome and employment status.

DETAILED DESCRIPTION:
Background: With an incidence of 6 in 1000 live born children congenital heart disease is among the most common birth defects. Survival rates of children with CHD have significantly improved during the past decades due to better surgical and intensive care medicine. Nowadays, even children requiring open- heart surgery for CHD most frequently have a good cardiac outcome and survive into adulthood. Even those with the most complex forms of CHD have sufficient cardiac outcome. However, impaired quality of life, mental health and behavior problems, as well as neurocognitive and motor impairments have been described to occur more frequently in children with CHD compared to healthy children and may persist into adolescence.

Current findings on QoL, psychological adjustment, and academic achievements in young adults with CHD are currently quite inconsistent due to methodological reasons. Moreover, little is known on risk factors for a negative outcome. To date, mainly medical risk factors have been examined while psychosocial characteristics (e.g., socioeconomic status, parenting, family characteristics) have not been systematically studied. Importantly, little is known about academic achievements and employment situations of young adults with CHD.

Aims: In this study the investigators aim to evaluate the psychosocial situation of adult CHD patients in terms of health-related quality of life, mental health, academic achievement, and employment status.

Methods: The study is designed as a case-control study beeing a mono-center project. The patient group will consist of a maximum of 350 patients with congenital heart disease treated at the cardiologic department of the University Hospital Zurich and a control group consisting of the same amount of also up to 350 individuals beeing good friends of the patients with same gender and similar age.

Recruitment: Participants will be consecutively recruited from May 1st, 2015 to April 30th, 2016. Eligible patients will be contacted by the study nurse during the outpatient consultation at the university hospital. Patients will be informed about the study during their consultation by the study nurse as well as the doctor with whom they have their appointment.The control group will be recruited as good friends (same gender, approx. same age) of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Congenital heart disease (Tetralogy of Fallot, Transposition of the great arteries, univentricular heart disease, ventricular septal defect) treated at the University hospital Zurich.
* Male and Female subjects 18 years to 30 years of age
* Written informed consent by the participant after information about the project
* In command of the German language

Exclusion Criteria:

* Diagnosis of a chromosomal or genetic syndrome as well as other congenital or acquired neurological impairments leading to mental disorders

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Yound adult patients with congenital heart disease
Sampling Method: Non-Probability Sample
Enrollment: 325 (Actual)
Dates: Start 2015-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Health related Quality of life | up to 12 months
  Health related Quality of life will be assessed by the SF-36 questionnaire (Bullinger & Kirchberger, 1998).

SECONDARY OUTCOMES:
Psychological adjustment | up to 12 months
  Psychological adjustment will be assessed by the symptom checklist-27 (SCL-27).
Academic achievement / employment situation | up to 12 months
  Academic achievement / employment situation will be assessed by means of a self-developed questionnaire: Participants will be asked to give information on their own education by means of number of school years, number of school year repetitions, type of schooling, need for special schooling or tutoring, age at graduation from school, completed apprenticeship and current employment status.
Medical data | up to 12 months
  Medical data will be collected only for the patients from their medical records: Exact cardiac diagnosis, number of surgeries on cardio-pulmonary bypass, number of interventional procedures, current functional class (according to the New Your Heart Association functional class), biometric characteristics (body weight, height, body mass index), current clinical findings (oxygen saturation, respiratory rate, heart rate, blood pressure), current medication, previous cardiovascular complications (arrhythmias, heart failure, endocarditis, stroke), current echocardiographic findings (ventricular function, residual valve regurgitation or stenosis, residual shunts), data from exercise testing (maximal exercise capacity, maximal oxygen uptake, heart rate reserve), findings from cardiac catheterization and cardiac MRI or CT, if available.
Executive functions | up to 12 months
  Executive functions will be measured with the dysexecutive questionnaire (DEX) (Wilson, Alderman, Burgess, Emslie, & Evans, 1996).
Major life events | up to 12 months
  Major life events will be assessed for the previous 12 months by a 12-item scale regarding for example unemployment, change of domicile, death of family members or friends (Landolt & Vollrath, 1998).
Social support | up to 12 months
  Social support will be assessed by means of the the F-SozU, a 14-item short form questionnaire assessing subjectively perceived emotional and instrumental support as well as social integration (Fydrich, Sommer & Brähler, 2002).
Emotional regulation | up to 12 months
  Emotional regulation is measured with the FEEL-E, an inventory that assesses 12 strategies (6 adaptive, 6 maladaptive) for regulation of temper, fear and grief (Grob & Horowitz, 2014).
Socioeconomic status | up to 12 months
  Socioeconomic status will be calculated by means of a 6-point scale scoring for paternal occupation and maternal education.
Biographical information | up to 12 months
  Participants will be asked to give information on their family status, own children, citizenship, mother tongue and parents'mother tongue on the same questionnaire they fill out information about education and academic career.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Landolt, PHD, Principal Investigator — University Children's Hospital, Zurich
Locations (1):
- UniversityHospital Zurich, Zurich, Switzerland

REFERENCES:
- [Background] Bullinger, M. & Kirchberger, I. (1998). SF-36 Fragebogen zum Gesundheitszustand. Göttingen: Hogrefe.
- [Background] Burgess, P. W., Alderman, N., Wilson, B. A., Evans, J. J., & Emslie, H. (1996). The dysexecutive Questionnaire. In B. A. Wilson, N. Alderman, P. W. Burgess, H. Emslie, & J. J. Evans (Eds.), Behavioral assessment of the dysexecutive syndrome. Bury St. Edmunds, UK: Thames Valley Test Company.
- [Background] Landolt, M.A. & Vollrath, M.E. (1998). Life Event Scale. Zurich: University Children's Hospital.
- [Background] Fydrich, T., Sommer, G., & Brähler, E. (2007). Fragebogen zur sozialen Unterstützung (F-SozU). Göttingen: Hogrefe.
- [Background] Grob, A. & Horowitz, L.M., Fragebogen zur Erhebung der Emotionsregulation bei Erwachsenen (FEELE). (2010). Bern: Huber